CLINICAL TRIAL: NCT01626001
Title: An Imaging Study to Compare Methods to Reduce 4DCT Image Acquisition Artifacts
Brief Title: Imaging Study Compare 4DCT Image
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-0631; 1dp20D007044-01 (Other: NIH Director's New Innovator Award)
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-08

CONDITIONS: Esophagus Cancer; Lung Cancer
Keywords: Esophagus Cancer; Lung Cancer; 4-dimensional computed tomography; 4D CT
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Cohort of 18 subjects evaluated. Subject will receive 4DCT cine acquisition gated using a respiratory signal from real-time position management (RPM) gating system. Maximum number of allowable images that may be acquired increased from 3000 to 5999 images. Total imaging time for each subject < 60 minutes.
  Interventions: Procedure: 4D CT scans
- Cohort 2 (Experimental): Reproducibility of optimal 4DCT acquisition method determined from cohort 1 tested with cohort of 18 study subjects. Three 4DCT images acquired, all with acquisition method determined from cohort 1. Cohort also receives two spiral-mode 4DCT acquisitions.
  Interventions: Procedure: 4D CT scans

INTERVENTIONS:
Procedure: 4D CT scans — 4 (or 5 for Cohort 2) 4DCT scans performed. 1 scan performed while breath held for less than 20 seconds. CT scans take about 5 minutes each to complete.
  Other Names: CT; X-ray; Computed Tomography

SUMMARY:
The goal of this clinical research study is to learn about ways to possibly reduce scanning errors when using 4-dimensional computed tomography (4D CT) scans to check lung function in patients with esophageal or lung cancer.

DETAILED DESCRIPTION:
Study Procedure:

By using 4D CT scans, researchers can create images that show how air moves through the lungs. This new method to check lung function may make better images than the standard methods. Researchers will compare 4 images of how air moves through your lungs and 1 image while you hold your breath.

Study Groups:

If you are found to be eligible to take part in this study (if the screening test is applicable) and you agree to take part in this study, you will be enrolled in 1 of 2 study groups, depending on when you join the study. There will be up to 18 participants in each group. In the first group, researchers will test several different methods to create images of how air moves through the lungs. Researchers will then select the most successful methods from the first group and try to do them again with the second group.

Study Visits:

You will have up to two visits for this study. At these visits, you will have four 4DCT scans performed (for Group 1) or five scans (for Group 2) using both the 4DCT and spiral CT, while you are breathing normally. You will also have 1 scan while you hold your breath for less than 20 seconds. The CT scans will take about 5 minutes each to complete. If the spiral CT scans for Group 2 cannot be completed on the same day as the 4DCT scans, you will be asked for your willingness to return at a later day to complete these.

The 4D CT scan will cover the entire chest area using the standard dose of radiation. A 2-inch plastic box will be placed on top of your chest to track the motion of your chest while you breathe during each scan. Some parts of your chest will be scanned up to 2 more times based on your breathing.

The entire scanning session will take about 45 minutes to complete.

Length of Participation:

Your active participation on the study will be over when you have completed your study visit.

Follow-Up Phone Call:

Within 7 days after your last study visit, the study staff will call you to ask about any side effects you may be having. This call should last about 2 minutes.

If anything unusual is found in the imaging, your cancer doctor will be told so that you can receive follow-up.

This is an investigational study. The CT scans used in this study are delivered using FDA-approved and commercially available systems. Creating images of how air moves through the lungs from 4D CT scans is considered investigational.

Up to 36 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign consent for the study.
2. Patients with pathologic diagnosis of esophagus or lung cancer.
3. Patient who plan to receive radiation therapy treatment at MD Anderson.
4. Patient >/=18 years of age

Exclusion Criteria:

1. Presence of an implanted electronic device.
2. Women who are pregnant or lactating, due to possible adverse effects on the developing fetus or infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Patient Percentage with 4DCT Acquisition Artifacts | 1 day
  Primary statistical analysis is intra-subject comparison of artifacts versus acquisition methods. In cohort 1: 4DCT acquisition techniques consist of 1) baseline acquisition, 2) extended acquisition, 3) real-time acquisition gating, and 4) re-imaging of bad segments. An automated computer scoring system, as described by Han et al., will be implemented and validated using the first 5 cases. To quantify 4DCT image quality, number and anatomic misplacement distance of artifacts will be measured, for each set of acquisition methods and each subject.

SECONDARY OUTCOMES:
Artifact Reproducibility Reducing 4DCT Acquisition | 1 day
  Winning acquisition method with lowest average misplacement per subject selected for evaluation of reproducibility. Goal is to quantify intra-subject variance for selected winning 4DCT acquisition method on image parameters significant for calculation of 4DCT ventilation images. Both acquisition artifacts and physiological parameters (global average HU, ΔHU, the tidal volumes, and the lung mass) assessed for reproducibility with evaluation of mean and variance.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guerrero, MD,PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org